CLINICAL TRIAL: NCT04809922
Title: Accuracy of Cardiac Wearables Devices to Detect Atrial Fibrillation in a Real-World Cohort of Patients; BASEL Wearable Study
Brief Title: Accuracy of Cardiac Wearables Devices to Detect Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-02425; kt21Badertscher
Record Dates: First submitted 2021-03-18; First posted 2021-03-22 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Atrial Fibrillation (AF)
Keywords: Cardiac Wearables Devices; Sinus rhythm (SR); Lead-intelligent Electrocardiogram (iECG); heart rhythm device accuracy
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: cardiac wearable devices — five cardiac wearable devices
  * Apple Watch, Apple Inc., Model Number: A1977 / A1978
  * Kardia Mobile, AliveCor Inc., AC-009/Kardia Mobile 6L, AliveCor Inc., AC-019
  * Fitbit Sense, Fitbit, Inc, Model Number: FB512
  * Samsung Galaxy Watch 3 Samsung Inc., Model Number: SM-R855F
  * Withings Scanwatch, Withings SA, Model Number: HWA09 Used for recording of one single-lead ECG. The results will be 274 compared to a simultaneous 12-lead ECG, which is considered the gold standard for detecting AF. There is no comparator in this trial.

SUMMARY:
Atrial fibrillation (AF) is the most common cardiac arrhythmia. This study is to assess the heart rhythm device accuracy of five cardiac wearable devices (Apple Watch, Kardia Mobile/Kardia Mobile 6L, Fitbit Sense, Samsung Galaxy Watch 3 and Withings Scanwatch, Withings SA, Model Number: HWA09) and its detection algorithms in identifying AF compared to a nearly simultaneously acquired physician-interpreted 12-lead ECG in a real world cohort of patients.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients undergoing electrophysiological study, pacemaker or implantable defibrillator (ICD) implantation or electric cardioversion at the University Hospital Basel are eligible for study participation and will be asked to participate

Exclusion Criteria:

* Use of a radial artery graft for coronary artery bypass grafting
* Tattoos located on the skin of the wrist or forearm where wearable device will be placed
* Patients receiving hemodialysis through arteriovenous fistula in the upper extremities
* Patients with inability to communicate and comply with all study requirements
* Patients who refused to participate in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing electrophysiological study, pacemaker or implantable defibrillator (ICD) implantation or electric cardioversion at the University Hospital Basel.
Sampling Method: Probability Sample
Enrollment: 312 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Heart rhythm device accuracy of cardiac wearable devices | one time assessment at baseline
  Heart rhythm device accuracy of five cardiac wearable devices (Apple Watch, Kardia Mobile/Kardia Mobile 6L, Fitbit Sense, Samsung Galaxy Watch 3 and Withings Scanwatch Withings SA, Model Number: HWA09) in detecting AF compared to nearly simultaneously acquired physician interpreted 12-lead ECG.
Heart rhythm device accuracy of physician-interpreted iECG | one time assessment at baseline
  Heart rhythm device accuracy of physician-interpreted iECG from a wearable device in detecting AF or SR compared to physician-interpreted 12-lead ECG

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Badertscher, Dr. med., Principal Investigator — Department of Cardiology, University Hospital Basel
Locations (1):
- Department of Cardiology, University Hospital Basel, Basel, Switzerland